CLINICAL TRIAL: NCT02439424
Title: The Effect of Reactive ATP™ on the Burden of Atrial Fibrillation in ICD Patients: The REACT-ICD Trial
Brief Title: The REACT-ICD Trial
Acronym: REACT-ICD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HHC-2015-0024
Record Dates: First submitted 2015-04-21; First posted 2015-05-08 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Atrial Tachyarrhythmia; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reactive ATP (Experimental): all enrolled subjects will have the Reactive ATP feature in their ICD turned "on"
  Interventions: Device: Reactive ATP

INTERVENTIONS:
Device: Reactive ATP — Reactive ATP turned to "on"

SUMMARY:
Recent advancements with implantable cardiac device technology include extensive diagnostic and therapeutic algorithms for prevention as well as termination of atrial tachyarrhythmias (ATA). Preventive atrial pacing (PAP) and a novel atrial antitachycardia pacing algorithm (Reactive ATP™) in conjunction with managed ventricular pacing (MVP) recently has been shown to reduce progression to permanent atrial fibrillation (AF) in pacemaker patients with intact atriovenous (AV) conduction and a history of ATA. Whether the use of Reactive ATP™ for reducing AF burden extends to patients with an implantable cardioverter defibrillator (ICD), who typically have structural heart disease and heart hailure (HF), is unknown.

DETAILED DESCRIPTION:
Atrial tachyarrhythmias (ATA) and heart failure (HF), which are well-recognized causes of morbidity and mortality, are growing and concerning issues in our patient population. In patients implanted with a dual-chamber implantable cardioverter defibrillator (ICD), progression of paroxysmal to persistent or permanent atrial fibrillation (AF) has been documented. Because of the untoward consequences of AF, such as development/worsening of HF or thromboembolic events (stroke and myocardial infarction [MI]), prevention of permanent AF has the potential to improve quality of life, reduce hospitalizations, and decrease the complications associated with AF.

Recent advancements with implantable cardiac device technology include extensive diagnostic and therapeutic algorithms for prevention as well as termination of ATA. Preventive atrial pacing (PAP) and a novel atrial antitachycardia pacing algorithm (Reactive ATP™) in conjunction with managed ventricular pacing (MVP) recently has been shown to reduce progression to permanent AF in pacemaker patients with intact atriovenous (AV) conduction and a history of ATA. Results of that study suggested that Reactive ATP™ specifically was responsible for this effect. Whether the use of Reactive ATP™ for reducing AF burden extends to patients with an implantable cardioverter defibrillator (ICD), who typically have structural heart disease and HF, is unknown.

The aim of this study is to evaluate the effectiveness of atrial antitachycardia pacing (Reactive ATP) in patients implanted with either a dual-chamber or cardiac resynchronization therapy (CRT) ICD who have a history of ATA.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients
* ≥18 years old (no upper age limit)
* previously implanted with a Medtronic dual-chamber or CRT ICD with capability of atrial antitachycardia pacing; specifically, Reactive ATP™ at least 9 months previously (six months data collection and implant occurring at least 3 months previously to allow healing and establishment of stable sensing)
* measured P wave in sinus rhythm of at least 0.8 mV
* >=6 months AT/AF burden data available, either from CareLink® or in-office interrogation
* >=1.0% AT/AF burden (hours in atrial fibrillation/total hours monitored) in the last 6 months
* No change in antiarrhythmic drug therapy (Vaughan-Williams class I or III) in the last 6 months

Exclusion Criteria:

* Persistent or permanent AT/AF (AF burden >95%)
* Cardioversion for atrial fibrillation or atrial flutter within the last 6 months, either intentional or as a result of a tachyarrhythmia therapy
* Ablation for atrial fibrillation or atrial flutter within the last 9 months (6 months data collection following a 3 month blanking period post procedure)
* Reactive ATP™ previously programmed on
* Measured P waves in sinus rhythm consistently <0.8 mV on repeat measurements.
* Unresolved artifactual AT/AF detection due to far-field R wave or other oversensing
* Expected generator change or other device surgery within six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation burden | 6 months
  % of time in atrial fibrillation = time in atrial fibrillation (over 6 months of study) / 6 months

SECONDARY OUTCOMES:
Persistent/permanent atrial fibrillation | 6 months
  number/percentage of patients in persistent (7 days) or permanent atrial fibrillation
cardioversion | 6 months
  number/percentage of patients who underwent cardioversion
cardiovascular hospitalization | 6 months
  number/percentage of patients who were hospitalized for cardiac-related issues
percentage of ventricular pacing | 6 months
  percentage of ventricular beats that are paced by the ICD
Ventricular tachycardia/Ventricular fibribilation ICD therapies | 6 months
  number of appropriate or inappropriate therapies (ATP [antitachycardiac pacing] or shock)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Zweibel, MD, Principal Investigator — Hartford HealthCare
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Background] Swerdlow CD, Schsls W, Dijkman B, Jung W, Sheth NV, Olson WH, Gunderson BD. Detection of atrial fibrillation and flutter by a dual-chamber implantable cardioverter-defibrillator. For the Worldwide Jewel AF Investigators. Circulation. 2000 Feb 29;101(8):878-85. doi: 10.1161/01.cir.101.8.878. PMID 10694527
- [Background] Lampe B, Hammerstingl C, Schwab JO, Mellert F, Stoffel-Wagner B, Grigull A, Fimmers R, Maisch B, Nickenig G, Lewalter T, Yang A. Adverse effects of permanent atrial fibrillation on heart failure in patients with preserved left ventricular function and chronic right apical pacing for complete heart block. Clin Res Cardiol. 2012 Oct;101(10):829-36. doi: 10.1007/s00392-012-0468-7. Epub 2012 May 16. PMID 22588842
- [Background] Israel CW, Gronefeld G, Ehrlich JR, Li YG, Hohnloser SH. Long-term risk of recurrent atrial fibrillation as documented by an implantable monitoring device: implications for optimal patient care. J Am Coll Cardiol. 2004 Jan 7;43(1):47-52. doi: 10.1016/j.jacc.2003.08.027. PMID 14715182
- [Background] Boriani G, Padeletti L, Santini M, Gulizia M, Capucci A, Botto G, Ricci R, Molon G, Accogli M, Vicentini A, Biffi M, Vimercati M, Grammatico A. Predictors of atrial antitachycardia pacing efficacy in patients affected by brady-tachy form of sick sinus syndrome and implanted with a DDDRP device. J Cardiovasc Electrophysiol. 2005 Jul;16(7):714-23. doi: 10.1111/j.1540-8167.2005.40716.x. PMID 16050828
- [Background] Israel CW, Ehrlich JR, Gronefeld G, Klesius A, Lawo T, Lemke B, Hohnloser SH. Prevalence, characteristics and clinical implications of regular atrial tachyarrhythmias in patients with atrial fibrillation: insights from a study using a new implantable device. J Am Coll Cardiol. 2001 Aug;38(2):355-63. doi: 10.1016/s0735-1097(01)01351-1. PMID 11499724